CLINICAL TRIAL: NCT03819608
Title: Neuromodulation and Neurorehabilitation for Treatment of Functional Deficits After mTBI and PTSD
Brief Title: Neuromodulation and Neurorehabilitation for mTBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Theresa Pape, Research Health Scientist, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 1034818
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Mild Traumatic Brain Injury; Post Traumatic Stress Disorder
Keywords: mTBI; PTSD; intermittent theta burst stimulation; cognitive training; neuroimaging
MeSH Terms: conditions — Brain Concussion; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- real APT+ real iTBS (Experimental): real APT+ real iTBS included 30 1-hour treatment sessions will be provided 3/week. Sessions will be conducted for 10 weeks. APT-III is a computer based cognitive training program. iTMS will be applied at 5Hz rate; each burst consists of 3 pulses delivered at 50Hz rate. The bursts are applied for 2s with 8s inter-burst-intervals, for a total of 600 pulses. The total stimulation time per session is approximately 192s (~ 3 minutes). Participants randomized to active iTBS will receive stimulation at the right dorsolateral prefrontal cortex at 80% active motor threshold .
  Interventions: Device: real iTBS; Behavioral: real APT
- real APT + placebo iTBS (Active Comparator): 30 1-hour treatment sessions will be provided 3/week. Sessions will be conducted for 10 weeks. APT-III is a computer based cognitive training program. Participants randomized to placebo iTBS will not receive any iTBS stimulation.
  Interventions: Behavioral: real APT; Device: placebo iTBS
- placebo APT+ real iTBS (Active Comparator): 30 1-hour treatment sessions will be provided 3/week. Sessions will be conducted for 10 weeks. Placebo APT-III is a computer based active control cognitive training program. Bursts of TMS pulses will be applied at 5Hz rate; each burst consists of 3 pulses delivered at 50Hz rate. The bursts are applied for 2s with 8s inter-burst-intervals, for a total of 600 pulses. The total stimulation time per session is approximately 192s (~ 3 minutes). Participants randomized to active iTBS will receive stimulation at the right DLPFC at 80% active motor threshold .
  Interventions: Device: real iTBS; Behavioral: placebo APT
- placebo APT+ placebo iTBS (Active Comparator): 30 1-hour treatment sessions will be provided 3/week. Sessions will be conducted for 10 weeks. Placebo APT-III is a computer based active control cognitive training program. Participants randomized to placebo iTBS will not receive any iTBS stimulation.
  Interventions: Behavioral: placebo APT; Device: placebo iTBS

INTERVENTIONS:
Device: real iTBS — Intermittent Theta Burst Stimulation (iTBS) is a form of repetitive transcranial magnetic stimulation (rTMS), which uses short magnetic field pulses applied to the scalp to induce currents in the underlying brain. iTBS will be delivered with the Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P. The Magpro Cool Coil B65 A/P can be switched to active or placebo (A/P).
  Other Names: intermittent Theta Burst Stimulation
  Arms: placebo APT+ real iTBS; real APT+ real iTBS
Behavioral: real APT — APT-III is an attention processing training program
  Other Names: Attention Processing Training-III
  Arms: real APT + placebo iTBS; real APT+ real iTBS
Behavioral: placebo APT — computerized cognitive training
  Other Names: Active Control APT
  Arms: placebo APT+ placebo iTBS; placebo APT+ real iTBS
Device: placebo iTBS — delivered with the Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P. The Magpro Cool Coil B65 A/P can be switched to active or placebo (A/P).
  Other Names: sham intermittent Theta Burst Stimulation
  Arms: placebo APT+ placebo iTBS; real APT + placebo iTBS

SUMMARY:
This study will determine (i) the magnitude of immediate and sustained effects of a current clinical standard interactive computer attention processing training (APT) when combined with intermittent theta burst stimulation (iTBS), a type of repetitive transcranial magnetic stimulation and (ii) determine how APT + iTBS changes the neurocognitive system of attention in individuals with persistent attention deficits related to mTBI +/- PTSD.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and no older than 80 years of age
* 3 months post exposure to mTBI event
* Have a history of mTBI with PTSD OR mTBI without PTSD as defined by formalized measures to classify mTBI based on the Symptom Attribution and Classification Algorithm (SACA) and the PTSD Module L of the SCID
* Endorse at least moderate severity on at least one of the four cognitive complaints in the Neurobehavioral Symptom Inventory

Exclusion Criteria:

* Participating in another research study
* Non-fluent in English (speaking and reading)
* History of epilepsy pre-injury
* Receiving antiepileptic treatment for documented active seizures in the past 6 months
* Taking medications that lower seizure threshold including antipsychotics, trazodone and tramadol
* History of surgery on blood vessels in brain and/or valves of the heart
* History of brain hemorrhage, neurovascular conditions and neurodegenerative disorders
* History or current diagnosis of psychotic spectrum disorders (i.e. bipolar, schizophrenia)
* Significant heart disease as determined by physician review of medical chart
* Pregnant at time of enrollment or any time during study participation
* MRI or TMS/iTBS contraindications such as claustrophobia, metal in eyes/face or brain
* Cardiac pacemakers/defibrillators, cochlear implants, nerve stimulators, intracranial metal clips
* Diagnosis of moderate or severe TBI (loss of consciousness > 30 minutes, alteration of consciousness > 24 hours, post traumatic amnesia or neuropsychological testing results
* Prescribed dosage of mental health medications have been altered within the month preceding study screening. Any participant whose mental health medication(s) has/have changed, within 30 days of study screening. The following are considered a medication change: the addition of or discontinuation of medication, a change in the dose or dosage (daily amount) of medication.
* Taking prescribed CNS stimulants and choosing to not stop these medications during study participation
* Taking prescribed CNS stimulants and choosing to not stop these medications during study participation
* Testing positive for opiates and do not have a prescription for opiates. If on prescription opiates and taking more than the equivalent of 200 mg of morphine per day.
* Questionably valid test performance as indicated by a score of ≤ 85% on the Immediate Recognition, Delayed Recognition or Consistency Scales of the Medical Symptom Validity Test (MSVT) and clinical determination of questionable performance validity by a neuropsychologist on the research team
* Actively suicidal as evidenced by plan to harm or recent attempt communicated on the Structured Clinical Interview for DSM-V (SCID-5).
* Increased Intracranial Pressure (ICP) as evidenced through a funduscopic evaluation or on the baseline MRI scan.
* Moderate or severe cannabis use disorder defined by ≥ 4 symptoms on the SCID-5
* Severe alcohol use disorder defined by ≥ 6 symptoms on the SCID-5
* Baseline systolic BP greater or equal to 170

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Mayo Portland Adaptability Inventory (MPAI) | baseline, 5 weeks, 10 weeks, 20 weeks
  Self-reported ability, adjustment and community participation. It is comprised of 30 items and three subscales: Ability Index, Adjustment Index and Participation Index. Items are scored on a 5-point Likert scale, with lower scores indicating higher levels of functioning.

SECONDARY OUTCOMES:
change in the PTSD Checklist (PCL) | baseline, 5 weeks, 10 weeks, 20 weeks
  20-item self-report measure assessing the distress associated with PTSD symptoms. The higher the score, the worse the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa LB Pape, Dr.PH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Moody Neurorehabilitation Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
FITBIR